CLINICAL TRIAL: NCT06493214
Title: Utilizing a SMART Intervention Design to Optimize Participant Adherence in Home-based Behavioral Interventions
Brief Title: Interrupting Prolonged Sitting With ACTivity (InPACT) at Home Optimization Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Rebecca Hasson, Associate Professor, University of Michigan
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HUM00253411
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-08

CONDITIONS: Adherence, Treatment; Physical Inactivity
MeSH Terms: conditions — Treatment Adherence and Compliance; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: In Stage 1 of the intervention, 30 child participants will enroll in the InPACT at Home exercise program, aiming to complete three 8-minute videos per day, five days a week. After four weeks, response rates will be evaluated. In Stage 2, ten participants will continue the program, while the other 20 will receive additional support via daily text messages or personalized activity calendars. In Stage 3, participants will be re-randomized to receive further support through either Tailoring or Coaching, with feasibility and response rates assessed throughout the 60-day study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Calendars + Pings + Coaching (Experimental): Intervention is administered online (electronic calendars and text message pings) and virtually (coaching).
  Interventions: Behavioral: Physical activity
- Calendars + Pings + Tailored Calendar (Experimental): Intervention is administered online (electronic calendars and text message pings).
  Interventions: Behavioral: Physical activity
- Calendars + Pings + Pings (Experimental): Intervention is administered online (electronic calendars and text message pings).
  Interventions: Behavioral: Physical activity
- Calendar + Tailored calendars + Pings (Experimental): Intervention is administered online (electronic calendars and text message pings).
  Interventions: Behavioral: Physical activity
- Calendar + Tailored calendars + Coaching (Experimental): Intervention is administered online (electronic calendars) and virtually (coaching).
  Interventions: Behavioral: Physical activity
- Calendar + Tailored calendars (Experimental): Intervention is administered online (electronic calendars).
  Interventions: Behavioral: Physical activity
- Calendars + Pings (Experimental): Intervention is administered online (electronic calendars and text message pings).
  Interventions: Behavioral: Physical activity
- Calendars + Tailored calendar (Experimental): Intervention is administered online (electronic calendars).
  Interventions: Behavioral: Physical activity
- Calendars (Experimental): Intervention is administered online (electronic calendars).
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — Participants will be asked to complete three eight-minute InPACT at Home exercise videos per day, five days a week, for 12 weeks.

SUMMARY:
Adherence refers to how well a person follows a recommended and agreed-upon course of action. Adherence is necessary for desired clinical outcomes and can include attending appointments, making lifestyle changes, and following home-based regimens for themselves or someone for whom they care for. Adherence to home exercise programs can be as low as 50%, directly impacting program effectiveness. There are many reasons why an individual may struggle to adhere, which may include perceived barriers such as not having enough time, reduced self-efficacy, the belief that the program is ineffective, or seeing early positive results so they then feel they do not need to continue with the program. For children, low skill level and lack of parental support are additional barriers to program adherence. A Sequential Multiple Assignment Randomized Trial (SMART) intervention is an intervention design that guides the adaptation of treatments over time. Adaptation refers to the use of dynamic information about a person (or family) to decide whether and how to intervene. SMART interventions are intended to address the unique and changing needs of individuals. The proposed study will examine the feasibility of using a 12-week (60-day) adaptive intervention design to optimize child adherence to a home exercise program. To advance equitable adherence to home exercise programs, there is a pressing need to develop strategies that support all children and families. The proposed study will provide new knowledge regarding the utility of adaptive interventions to optimize participation engagement in behavioral interventions in community contexts.

DETAILED DESCRIPTION:
Experimental protocol: In Stage 1 of the intervention, 30 child participants will enroll in a home exercise program called InPACT at Home. The objective is for each participant to complete three 8-minute exercise videos per day, five days a week (30-45 minutes total daily). Participants will receive a calendar with links to the daily videos on a private YouTube channel. The response rate will be evaluated at the end of week 4, consistent with the original InPACT at Home pilot feasibility trial timeframe. Participants who do not complete Stage 1 will still be eligible to participate in Stage 2, focusing on adherence. Stage 2 involves ten participants continuing with InPACT at Home, while the remaining 20 will be randomly assigned to additional support groups. These groups include daily text message reminders (pings) for ten participants and personalized activity calendars based on individual physical activity preferences for the other ten. The response rate will again be assessed at the end of week 8. In Stage 3, seven participants initially assigned to InPACT at Home + Pings will be randomly reassigned to receive further support through either Tailoring (Condition A) or Coaching (Condition B). Similarly, seven participants initially assigned to InPACT at Home + Tailoring will be re-randomized to receive additional support via either Pings (Condition D) or Coaching (Condition E). Seven participants initially receiving no support will be re-randomized to receive either Pings (Condition G) or Tailoring (Condition H). The primary objective of this pilot project is to assess the feasibility of the study design, ensuring that the response rate does not influence randomization. The study duration is 60 days.

Intervention Components: The InPACT at Home intervention consists of a structured calendar of activities and high-quality exercise videos. Additional supports include personalization of the activity calendar to individual preferences, daily text message reminders to parents, and coaching sessions aimed at overcoming household barriers to participation. Previous research has validated the feasibility of InPACT at Home, while other studies support the effectiveness of the chosen support mechanisms.

Measurements: Consented participants will undergo pre- and post-intervention assessments including physical activity enjoyment, habitual physical activity levels, anxiety and depression symptoms, emotion regulation, and parent support for physical activity. These measures will inform a larger SMART study evaluating the impact of InPACT at Home on child social-emotional health.

Measurement Tools:

* Physical Activity Enjoyment Scale: A validated questionnaire assessing enjoyment during physical activity.
* Physical Activity Questionnaire for Children (PAQ-C): Assesses pre- and post-intervention physical activity levels.
* Patient Health Questionnaire-9 (PHQ-9) and General Anxiety Disorder-7 (GAD-7): Measure depression and anxiety symptoms, respectively.
* Difficulties in Emotion Regulation Scale-Short Form: Evaluates emotion regulation abilities.
* Parental Support of Physical Activity Questionnaire: Assesses parental support for child physical activity.
* Ratings of Perceived Exertion Scale: Measures perceived exertion during exercise sessions using a 10-point scale.

Measurements taken during the Experimental Conditions:

Feasibility will be determined by attrition rates and adherence to the intervention. Attrition will track participants who drop out, while dose will monitor those completing at least 40 of the 60 exercise videos. Video completion will be recorded on activity calendars signed off by parents, and view duration will be assessed using YouTube analytics. Objective physical activity data will be collected using FitBit monitors worn during activity breaks.

Statistical Considerations: Sample size for this pilot study is based on current budgetary constraints (n=30). Data from this study will generate pilot data to calculate effect sizes for a larger trial examining adherence and program effectiveness.

ELIGIBILITY:
Inclusion Criteria:

This study will include both males and females aged 8 to 12 years and their parent/guardian from various locations in Michigan. The investigators have chosen this age group because this is a critical age with physical activity participation declines (75% from the age of 9 to 15 years). To be included in the study, participants must:

1. Have access to a computer and internet at home.
2. Be proficient in English.

Exclusion Criteria:

Children will not be eligible for the study if they meet any of the following conditions:

1. Currently taking medications (e.g., iron, metformin, chemotherapeutic agents) that could impact their ability to engage in physical activity.
2. Previously diagnosed with conditions that could impact their ability to engage in physical exercise (e.g., uncontrolled asthma).
3. Answering "YES" to any question on the Physical Activity Readiness Questionnaire (PAR-Q)22 indicating the participant has a heart condition, high BP, experienced chest pains or dizziness during daily activities, or require a doctor's recommendation for supervision during exercise.
4. Diagnosed with a physical or mental disability that would make it difficult to answer questions or follow directions without the help of an adult.
5. Parent or caregiver has a physical or mental disability that would make it difficult for them to answer questions or assist their child with project-related activities, such as completing questionnaires in the laboratory.
6. Potential participants who are ineligible will be told so on their screening call and will not be enrolled.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Dose of exercise received | Mid-treatment (4 and 8 weeks), immediately post-treatment
  Dose will be measured by identifying the number of participants who complete 40 or more of the 60 videos (averaging 2 videos per day). The self-reported average number of total videos completed over the 60-day intervention will be recorded on the activity calendar sheets. To ensure accuracy, parents will sign off on the logs at the end of each week. Like other studies, video view duration will be assessed using YouTube analytics. To validate child physical activity, child participants will be requested to wear a physical activity wrist monitor (FitBit) during each activity break. This objective measure aims to confirm the level of activity during the video sessions. Established procedures for device placement, initialization, and processing, which have undergone validation, will be strictly adhered to during this process.

SECONDARY OUTCOMES:
Attrition | Mid-treatment (4 and 8 weeks), immediately post-treatment
  Attrition will be determined by calculating the total number of participants who drop out.
Dose of intervention supports received | Mid-treatment (4 and 8 weeks), immediately post-treatment
  Dose of intervention supports will be quantified as attendance at weekly coaching sessions (coaching) and text message reads (pings) throughout the intervention period31. Research staff will document dose.

OTHER OUTCOMES:
Physical activity enjoyment scale | baseline, 1-week post-treatment
  Enjoyment will be assessed using the Physical Activity Enjoyment Scale (PACES) questionnaire. Participants will be asked to reflect on how they felt about the exercises. Example questions include the following: "When I was active . . . I enjoyed it, When I was active . . . I felt bored; When I was active . . . it frustrated me." The scale is a combination of 16 positive and negative statements. The responses are scored on a 5-point Likert scale, 1 (disagree a lot) to 5 (agree a lot). Seven of the 16 statements were reverse coded. An enjoyment score is calculated by averaging the scores. The revised Physical Activity Enjoyment Scale has been validated in children and demonstrated high reliability in the present analysis (Cronbach alpha= 0.91). The scale ranges from 0 to 48. PACES scores below 24 are interpreted as lower enjoyment while being physically active.
Physical activity questionnaire for children | baseline, 1-week post-treatment
  Pre- and post- physical activity levels will be assessed using the Physical Activity Questionnaire for Children (PAQ-C). Questionnaire items are scored (range 1 to 5) and a score of 1 indicated low physical activity and a score of 5 indicated high physical activity. This questionnaire has been validated for children ages 7-14 years old of all races.
Anxiety symptoms | baseline, 1-week post-treatment
  Anxiety symptoms will be assessed using the General Anxiety Disorder-7 (GAD-7). GAD-7 consists of seven items measuring worry and anxiety symptoms. Each item is scored on a four-point Likert scale (0-3) with total scores ranging from 0 to 21; higher scores reflecting greater anxiety severity. Scores above 10 are in the clinical range The GAD-7 has shown good reliability and construct validity.
Depression symptoms | baseline, 1-week post-treatment
  Depression symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9). PHQ-9 consists of nine items measuring depressive symptoms corresponding to the diagnostic criteria for major depressive disorder. Each item is scored on a four-point Likert scale (0-3) with scores ranging from 0 to 27, with higher scores reflecting greater depression severity. Scores above 10 are in the clinically depressed range. PHQ-9 has shown good psychometric properties.
Difficulties with emotion regulation | baseline, 1-week post-treatment
  To assess emotion regulation, the investigators will employ the Difficulties in Emotion Regulation Scale-Short Form, which comprises 18 items. These items gauge various aspects of emotion regulation, including one's ability to accept emotional responses, engage in purposeful actions, control impulses, be aware of emotions, access emotion regulation strategies, and attain emotional clarity. Each item is rated on a five-point Likert scale, with scores ranging from 1 to 5, resulting in total scores that fall between 18 and 90. Higher scores suggest greater problems with emotion regulation. This instrument has been rigorously tested and confirmed to be reliable in both adolescent and adult populations.
Parent physical activity social support | baseline, 1-week post-treatment
  Parent physical activity support will be measured via the Activity Support Scale for Multiple Groups (ACTS-MG) survey, which is a 12-item questionnaire that assesses parental support for exercise and consists of four subscales representing logistic support (e.g., I take my child to places where he/she can be active), modeling (e.g., I encourage my child to be physically active by leading by example), use of community resources (e.g., I encourage my child to use resources in our neighborhood to be active), and limiting sedentary activities (e.g., I limit how long my child plays video games). Items are scored on a 4-point Likert-type scale ranging from 1 (strongly disagree) to 4 (strongly agree), with higher scores indicating greater parental support for physical activity.
Rating of perceived exertion | during treatment
  Perceived exertion during each exercise condition, the Ratings of Perceived Exertion (RPE) scale for children will be used (Borg 1998). At the completion of each exercise video, participants look to the RPE scale and answer the question, "How hard do you feel you are working?" Participants will respond by selecting a number on a 10-point scale that reflects their perceived exertion (1= "Very, very easy" to 10 = "So hard, I'm going to stop"). The RPE scale has been validated in children.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Hasson, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
For the proposed research, the investigators will enroll 30 children. The investigators will be collecting physical activity and questionnaire data from these participants. All data will be de-identified. The investigators do not anticipate sharing data or samples with other investigators, but the investigators will make data available for sharing with other researchers if they sign a data sharing agreement indicating that:
  1. They will use the data for research purposes only.
  2. All data will be retained on a secure/password protected computer and computer program.
  3. If the identity of any participant is compromised, they will inform us immediately.
  4. Commitment to destroy or return the data after their analysis is complete

DOCUMENTS (2):
  • Informed Consent Form: Informed Consent Form (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT06493214/ICF_000.pdf
  • Informed Consent Form: Informed Assent Form (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/14/NCT06493214/ICF_001.pdf